CLINICAL TRIAL: NCT01974648
Title: ED 50 of Propofol for Supreme LMA Insertion With and Without Remifentanil. A Randomized Trial
Brief Title: Propofol for Supreme LMA Insertion With and Without Remifentanil
Acronym: SC50
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: FIBHGMECNC002-2011
Record Dates: First submitted 2013-10-21; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Patients Requiring Ambulatory Surgery Under General Anesthesia
Keywords: Laryngeal Mask Airway Supreme; propofol; remifentanil; effective dose of intravenous propofol; ED50
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Active Comparator): In control group, propofol concentrations will start at 4 μg ml-1, with 0,5 μg ml-1 as the step size, with the coadministration of saline.
  Interventions: Drug: propofol
- propofol and remifentanil (Experimental): In propofol-remifentanil group, propofol + remifentanil at a target-controlled infusion 5 ng/mL will be coadministered.
  Interventions: Drug: propofol and remifentanil

INTERVENTIONS:
Drug: propofol
  Arms: propofol
Drug: propofol and remifentanil
  Arms: propofol and remifentanil

SUMMARY:
The aims of this study were to determine the clinically required concentration of propofol for LMA Supreme insertion, and to examine to what extent remifentanil reduces the dose of propofol and improves conditions for it's insertion.

DETAILED DESCRIPTION:
The single-use Laryngeal Mask Airway SupremeTM (SLMA, Laryngeal Mask Company Limited, Singapore) is a new single use supraglottic airway device introduced recently that present combined features of the LMA ProSealTM (PLMA, Laryngeal Mask Company Limited) and the LMA FastrachTM (FLMA, Laryngeal Mask Company Limited). The mask has an anatomically shaped airway tube, elliptical in cross-section that facilitates easy insertion and minimizes accidental rotation. The cuff bowl is designed to prevent airway kinking and offer higher airway seal pressures around the laryngeal opening than the LMA ClassicTM (CLMA, Laryngeal Mask Company Limited) It has a drain tube that provides functional separation of the respiratory and digestive tracts to prevent gastric aspiration. Even though insertion of the SLMA is associated with a higher initial success rate, fewer airway manipulations and a safe and effective airway during anaesthesia, the anaesthetic techniques for its insertion were not standardised. Most available data on the requirements of anaesthetic drugs and co-induction agents used for insertion of SLMA originate from research involving other assessments of the SLMA such as the seal with respiratory and gastrointestinal tract.We tested for differences in the predicted concentration of propofol with and without remifentanil for insertion of the SLMA.

Methods: 50 patients ASA class I or II aged 18-75 years undergoing ambulatory elective surgery will be randomized to one of two groups: those who receive propofol + saline (control group: n = 25) or propofol + remifentanil (propofol-remifentanil group: n=25). We will use target-controled infusions (Alaris®PK) for both drugs: propofol (Marsh et al.´s pharmacokinetic model) and remifentanil (Minto et al.´s pharmacokinetic model). The patients wil be premedicated with midazolam 1 mg iv before surgery. The target concentration for each patient was determined using the Dixon´s up-and-down method. Predetermined propofol and remifentanil blood and effect site concentrations were held constant for at least 10 min. After equilibration of plasma and effect site propofol concentrations, the SLMA will be inserted, and secured according to the manufacture´s recommendations, without the use of muscle relaxants. In control group, propofol concentrations will start at 4 μg ml-1, with 0,5 μg ml-1 as the step size, with the coadministration of saline. In propofol-remifentanil group, propofol + remifentanil at a target-controlled infusion 5 ng/mL will be coadministered. A single measurement will be obtained from each patient. If the patient reacted with movement, the propofol concentration for the next patient was increased by 0.5 μg ml-1 ±1 ; if there was no movement, it was decreased by 0.5 μg ml-1 ±1 . Movement was defined as bucking or gross purposeful muscular movement within 1 min of LMA insertion. Values of Cp 50 wil be determined by calculating the midpoint concentration after at least seven crossover points (movement/non movement) will be obtained in each group.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-II patients Scheduled to ambulatory surgery Need of general anaesthesia General anaesthesia usually performed with laryngeal mask Negative pregnancy test in women. Signed informed consent.

Exclusion Criteria:

* Patients with a potentially difficult airway o (Mallampati III or IV, a limited mouth opening and/or cervical spine disease) Patients with reactive airway disease Signs of upper respiratory infection, Patients who had a risk of gastric aspiration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The concentration of propofol with and without remifentanil for insertion of the SLMA | at insertion of SLMA
  Comparison of he concentration of propofol with and without remifentanil for insertion of the SLMA

SECONDARY OUTCOMES:
changes in Systolic Blood Pressure, Diastolic Blood Pressure and Heart Rate | basal and every 3 minutes until 6 minutes after insertion of the SLMA
BIS | before and after SLMA insertion(every min until min 6)
  BIS data after SLMA insertion with both anaesthetic techniques
Fibrescope evaluation | after SLMA insertion
  Fibrescope evaluation of the SLMA Of the view of the glottis
blood pressure(Hypertension or hypotension) | before and after SLMA insertion(every min until min 6)
heart rate (tachycardia or bradycardia) | before and after SLMA insertion(every min until min 6)
  tachycardia or bradycardia requiring treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matilde Zaballos, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Marañon Servicio de Anestesiologia y Reanimación, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Zaballos M, Bastida E, Agusti S, Portas M, Jimenez C, Lopez-Gil M. Effect-site concentration of propofol required for LMA-Supreme insertion with and without remifentanil: a randomized controlled trial. BMC Anesthesiol. 2015 Oct 6;15:131. doi: 10.1186/s12871-015-0115-8. PMID 26438179